CLINICAL TRIAL: NCT04152278
Title: Chlamydia Tracomatis and Other Lower Genital Tract Infections Among Women With Unexplained Early Miscarriage
Status: Completed | Type: Observational
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Sahar MY Elbaradie, associate Professor, Fayoum University Hospital
Other Study IDs: fayoumUH
Record Dates: First submitted 2019-11-02; First posted 2019-11-05 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Early Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — cervicovaginal swabs, serum samples and placental tissues
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: The study group included 300 women presenting with unexplained spontaneous miscarriage or missed abortion during the first and early second trimester of pregnancy (8-16 weeks gestational age). The included women aged 18 to 45 years old.
  Interventions: Diagnostic Test: cervicovaginal culture and qPCR for chlamydial trachomatis and wadallia chondrophila
- control group: The control group included 300 women with normal pregnancy, recruited from women attending the antenatal clinic of gestational age 8-16 weeks. The included women aged 18 to 45 years old.
  Interventions: Diagnostic Test: cervicovaginal culture and qPCR for chlamydial trachomatis and wadallia chondrophila

INTERVENTIONS:
Diagnostic Test: cervicovaginal culture and qPCR for chlamydial trachomatis and wadallia chondrophila — three cervicovaginal swabs were obtained: one was used for a smear test of vaginal fluid pH evaluation and direct microscopy, the second swabs, cultured for aerobic and anaerobic bacteria and yeasts, the third was eluted in 2-sucrose-phosphate (2SP) based transport medium. Placental samples from the study group were cultured for aerobic and anaerobic bacteria. Placenta sample and 2SP medium were stored at -80°C until their analysis by real time PCR (qPCR)
  Other Names: placental culture and qPCR; study group only

SUMMARY:
Although one fourth of pregnant women experience at least 1 abortion, yet only 50% of causes are identified. Pregnancy loss can result from viral, bacterial, and other infections. It can reach the fetoplacental units through blood born or local spread. Lower genital tract infections- a potentially preventable infections- was suggested as a cause of spontaneous miscarriage. It was reported in 15 and 66% of early and late miscarriages respectively. These infections are also commonly encountered among apparently healthy looking pregnant women with an overall prevalence of 40-54%. If left untreated it can lead to premature rupture of the membranes, preterm birth, low birth weight, Fetal loss, neonatal ophthalmic and pulmonary damage.

DETAILED DESCRIPTION:
Abortion was defined by the World Health Organization and the National Center for Health Statistics as pregnancy termination before 20 weeks of gestational age or fetal weight smaller than 500 grams. Abortion is termed early or late if it occurs before 12 weeks or between 12 and 24 weeks of gestation respectively.

Spontaneous abortion prevalence is not exactly known as it varies according to the used method of identification. Wilcox and colleagues in 1988 reported a prevalence of 31 % of pregnancy loss after implantation and over 2/3 of them were clinically silent.

Although one fourth of pregnant women experience at least 1 abortion, yet only 50% of causes are identified. Pregnancy loss can result from viral, bacterial, and other infections. It can reach the fetoplacental units through blood born or local spread.

Lower genital tract infections- a potentially preventable infections- was suggested as a cause of spontaneous miscarriage. It was reported in 15 and 66% of early and late miscarriages respectively. These infections are also commonly encountered among apparently healthy looking pregnant women with an overall prevalence of 40-54%. If left untreated it can lead to premature rupture of the membranes, preterm birth, low birth weight, Fetal loss, neonatal ophthalmic and pulmonary damage.

The suggested mechanisms that genital tract infection can cause abortions are encountered are fetal or placental infection with production of toxic metabolites.

Some organisms like Brucella abortus, Campylobacter fetus, and Toxoplasma gondii can cause abortion in livestock. Their effects in human is unclear. Most infections were not linked to abortions except Chlamydia trachomatis, which was detected in 4% of abortuses compared with < 1 percent of controls.

Chlamydia trachomatis infection incidence was markedly increased in the last years and is responsible for many gynecological conditions as pelvic inflammatory disease and infertility and pregnancy complications as preterm birth and premature rupture of membranes but its relation to early pregnancy loss remains unrecognized.

Baud et al assumed an association between miscarriage and serologic/molecular evidence of C. trachomatis infection. This was evident by the higher prevalence of immunoglobulin G against C. trachomatis in the miscarriage group than in the control group (15.2% vs. 7.3%; p = 0.018) that remained significant after adjustment for age, origin, education, and number of sex partners (odds ratio 2.3, 95% confidence interval 1.1-4.9).

Polymicrobial infection was associated with 2 - 4fold increase in abortion. Data concerning a link between some other infections and increased abortion are conflicting. Oakeshott and coworkers (2002) reported an association between second-, but not first-, trimester miscarriage and bacterial vaginosis with a relative risk of miscarriage before 16 weeks' gestation of 1.2 (0.7 to 1.9).

The present study is designed to determine prevalence of genital tract infections and its relation to occurrence of early miscarriage in women with recent unexplained spontaneous miscarriages

ELIGIBILITY:
Inclusion Criteria:

* women with unexplained spontaneous miscarriage or missed abortion during the first and early second trimester of pregnancy (8-16 weeks gestational age).
* women with normal pregnancy, attending the antenatal clinic of gestational age 8-16 weeks.
* The included women aged 18 to 45 years old.

Exclusion Criteria:

* women with miscarriage at a gestational age of more than 18 weeks,
* those with documented causes of miscarriage as fetal or uterine anomalies, antiphospholipid syndrome or endocrine factors and
* women who received recent antibiotic, antifungal or antiprotozoal treatment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study group included 300 women presenting with unexplained spontaneous miscarriage. The control group included 300 women with normal pregnancy, recruited from women attending the antenatal clinic of gestational age 8-18 weeks.
  All participants were subjected to full history, careful general and abdominal examination, Cervicovaginal swabs, urine and blood sampling in addition to placental sampling from study group.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
the association of lower genital tract infection with spontaneous miscarriage | one year
  relation between genital tract infection and miscarriage

CONTACTS AND LOCATIONS:
Overall Officials: sahar MY Elbaradie, a.Professor, Principal Investigator — Fayoum University Hospital
Locations (1):
- sahar M.Y elbaradie, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided